CLINICAL TRIAL: NCT03714399
Title: A Prospective Observational Study Into Muscle Recovery Following Aortic Surgery Induced Intensive Care Unit-acquired Weakness (VARIANCE).
Brief Title: Muscle Recovery Following Aortic Surgery Induced ICUAW.
Acronym: VARIANCE
Status: Completed | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 012396 (VARIANCE)
Record Dates: First submitted 2018-06-05; First posted 2018-10-22 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2021-11

CONDITIONS: Aortic Diseases; Intensive Care Unit Syndrome; Intensive Care Neuropathy; Intensive Care (ICU) Myopathy; Critical Illness Myopathy; Surgery
Keywords: Intensive Care Unit Acquired Weakness (ICUAW); Critical Illness Polyneuromyopathy (CIPM); Health Related Quality of Life (HRQoL); Ultrasound (US); Cardiac Surgery; Rectus Femoris Cross Sectional Area (RFcsa)
MeSH Terms: conditions — Aortic Diseases; Muscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Muscle biopsies attained during surgery from the thigh and chest wall will undergo histological analysis. Blood samples (plasma and buffy coat) will also be analysed for mediators and markers of oxidative stress injury (e.g. 8-isoprostane), inflammation (e.g. GDF-15 and soluble tumour necrosis factor receptor) and injury to multiple organs will be quantified. Urine will be used to measure albumin-creatinine ratio (ACR) as a marker of endothelial injury.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICUAW group: The physical and psychological effects of ICUAW on patients undergoing aortic valvular surgery will be observed. Physical function and HRQoL will be analysed and correlated with RFcsa. Additionally, biological markers will be used to understand molecular and genomic profiles.

SUMMARY:
To identify determinants of 'good and bad recovery' from ICUAW and build knowledge around the timing of these processes. Also, the investigators want to discover the effects of ICUAW on physical function and HRQoL following aortic surgery.

DETAILED DESCRIPTION:
The aim is to identify determinants of recovery from intensive care unit-acquired weakness (ICUAW) and to discover the effects of ICUAW on physical function and health-related quality of life (HRQoL) after critical illness. This phenomenon has become more evident over recent years and still requires extensive research.

ICUAW is an umbrella term for more specifically, polyneuropathy and myopathy. Recent research has found that 50% of patients undergoing elective cardiac surgery lose significant muscle mass (9.6% in the wasters group) within the first seven days. These patients are receiving relatively uncomplicated surgery yet still suffering from muscle breakdown, which cannot be described by inactivity alone. ICUAW can lead to a significant increase in mortality, morbidity, hospital-acquired infections and pressure ulcers. Risk factors for ICUAW include neuromuscular blocking agents, hyperglycaemia, inactivity and sepsis. The correlation between a relatively homogenous (cardiac surgical) group and patient-centred outcomes during recovery such as functional ability and health-related quality of life (HRQoL) has been little studied.

Patients undergoing elective aortic valvular surgery at St Bartholomew's Hospital London will be recruited for the study. We have chosen the cardiac surgical model due to being a homogenous cohort where the time of insult from surgery from the cardiac bypass, can be measured in correlation with ICUAW. Due to the clamped aorta within the operation, prolonged periods of reduced blood flow to the body occurs, and therefore an element of ischaemia and reperfusion can lead to muscle wasting. Rectus Femoris cross-sectional area (RFcsa) will be measured at pre-determined intervals and the images then greyscaled and muscle quality assessed. To assess and quantify 'good and bad recovery,' we will correlate these tests with functional capacity and HRQoL. Additionally, Blood and urine samples will be taken at pre-defined intervals to observe for markers of oxidative stress, organ injury and molecular profiles. Muscle biopsies will be taken during surgery and observed for histological and fibre profiles.

The primary objective is to identify determinants of recovery from ICUAW and to discover the effects of ICUAW on physical function and health-related quality of life (HRQoL) after aortic valvular surgery. Specifically, to observe the cross-sectional area of the Rectus Femoris (RFcsa) and correlate this with muscle strength and HRQoL during the recovery phase. The RFcsa, hand-held dynamometry, knee straightening dynamometry, Free Fat Mass Index, standing and lying vital capacity and the short physical performance battery (SPPB) will be observed. Also, HRQoL will be measured using the reintegration to normal living index (RNLI), hospital and anxiety depression score (HADS), EQ-5D-5L (EuroQol research foundation). The primary endpoint will be once all these data are gathered and analysed.

The secondary aim is to understand the molecular and genomic profile of blood samples and the histology of the muscle biopsies. The secondary objective will be supported with additional data from urine analysis (Albumin-creatinine ratio, ACR). The secondary endpoint will be once these data are gathered and analysed.

ELIGIBILITY:
Inclusion Criteria:

* Above the age of 18
* Receiving elective aortic valvular surgery at Barts Health NHS Trust

Exclusion Criteria:

* Previous Stroke
* Neuromuscular disease
* Malignancy
* Underlying neuromuscular disease
* Paediatrics
* Non-consenting adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion criteria include any consenting adult receiving elective aortic surgery at Bartshealth NHS trust with no evidence of pre-hospital neuromuscular conditions.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-09-26 (Actual)

PRIMARY OUTCOMES:
To observe the change in cross sectional area of the Rectus Femoris (RFcsa) during critical illness and recovery. | Pre-operatively, day 7/Hospital Discharge and 6-15week follow up clinic.
  RFcsa will be calculated using B-mode ultrasound (US) at pre-determined time points. Additionally, the images acquired will have histogram analysis in adobe photoshop software. The RFcsa will be correlated with indices of muscle strength and HRQoL.
To Observe a change in Hand Held Dynamometry strength (grip strength) and correlate this with RFcsa, function and HRQoL during critical illness and recovery. | Pre-operatively, Day 7/Hospital Discharge and 6-15 week follow up clinic.
  Hand-held dynamometry will be calculated using the JAMAR hand-held hydraulic dynamometer. We will assess both hands and take the mean of 3 trials, producing a maximal grip result.
To observe a change in Knee straightening dynamometry, strength and joint moment (torque) and correlate this with RFcsa, function and HRQoL during critical illness and recovery. | Pre-operatively, Day 7/Hospital Discharge and 6-15 week follow up clinic.
  The test will be conducted using a Lafayette Manual Muscle Tester. Joint knee moment (torque) and strength will be measured.
To observe a change in Short Physical Performance Battery (SPPB) and correlate this with RFcsa, function and HRQoL during critical illness and recovery. | Pre-operatively, Day 7/Hospital Discharge and 6-15 week follow up clinic.
  SPPB will be measured at similar time points to understand a patients' functional status.
Lying and Standing Vital Capacity (FVC - forced vital capacity) and correlate this with RFcsa, function and HRQoL during critical illness and recovery. | Pre-operatively, Day 7/Hospital Discharge and 6-15 week follow up clinic.
  Lying and standing vital capacity will be measured using a hand held spirometer.
To measure Free Fat Mass Index (FFMI) and correlate this with RFcsa, function and HRQoL during critical illness and recovery. | Pre-operatively, Day 7/Hospital Discharge and 6-15 week follow up clinic.
  Free fat mass index (FFMI) and free fat mass (FFM) will be measured using the bodystat 1500 device. Other values will also be recorded from the test including body fat percentage and lean mass percentage. The body stat 1500 is an electrical device that uses electrical impedance to obtain results (objective data).
To measure the EQ-5D-5L (Euroscore) to assess general health and correlate this with the primary objective (RFcsa). | Pre operatively, Day 7/Hospital discharge and 6-15 week follow up.
  EQ5D-5L is a standardised tool that provides a simple generic measure of health. A summation of all the levels will be converted to a single index value using the EQ5D-5L crosswalk index value calculator. The general health score can range from 0 (worst health imaginable) to 100 (best health imaginable).
Hospital anxiety and depression score (HADS) to assess HRQoL and correlate this with the overall primary objective (RFcsa). | Pre-operatively, Day 7/Hospital discharge and 6-15 week follow up.
  The HADS is an assessment that measures whether a patients is suffering from anxiety or depression. HADS is a self assessment consisting of 16 items. A result of between 0 and 7 indicates a normal case, between 8 and 10 indicates borderline abnormal and between 11 and 21 indicates abnormal levels of anxiety and depression.
Reintegration to normal living index (RNLI) to assess HRQoL and correlate this with the overall primary objective (RFcsa). | Pre-operatively and 6-15 week follow up clinic.
  The RNLI is a 5 domain 11-tool item aimed at assessing the degree to which patients' who have experiences traumatic and incapacitating illness achieve reintegration into society. The RNLI score is based out of 110, which will be proportionally converted to create a score of 100. Zero indicates no integration whereas 100 implies full integration.

SECONDARY OUTCOMES:
The secondary aim is to understand the molecular profile (bloods). | Pre-operatively, Day 1, Day 3, Day 7/hospital discharge and 6-15 week follow up.
  Blood analysis will contain and analyse but not limited to markers of oxidative stress injury, inflammation, MiRNA and injury to multiple organs will be quantified. We will store Buffy coat and plasma to understand these profiles.
Urine Analysis | pre-operatively, Day 1, Day 3, Day 7/hospital discharge and 6-15 week follow up.
  Urine analysis observes albumin-creatinine ratio (ACR)
Muscle Biopsy | Intra-operatively
  A muscle biopsy will be taken from patients whilst under anaesthesia. The biopsy observes pathways relevant to muscle homeostasis using biochemical and molecular techniques.
Cardiac post operative morbidity score (C-POMS) will be used to calculate morbidity risk. | Day 3, day 5, day 8 and day 15 post cardiac surgery.
  C-POMS is additional data that will be collected and analysed. C-POMS is a validated tool assessing in-hospital morbidity burden (score 0-13) derived by noting the presence of 13 morbidity domains on days 3, 5, 8 and 15 after surgery. A higher score indicates a greater morbidity burden.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Grffiths, PhD FRCP, Principal Investigator — Substantive Employee and primary supervisor to PhD student; Julie Sanders, MSc, PhD, Principal Investigator — Director of research and supervisor to PhD student; Ashley Thomas, MSc, Principal Investigator — Substantive employee and PhD student
Locations (1):
- St Bartholomew's hospital (Barts NHS trust), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bloch SA, Donaldson AV, Lewis A, Banya WA, Polkey MI, Griffiths MJ, Kemp PR. MiR-181a: a potential biomarker of acute muscle wasting following elective high-risk cardiothoracic surgery. Crit Care. 2015 Apr 7;19(1):147. doi: 10.1186/s13054-015-0853-5. PMID 25888214